CLINICAL TRIAL: NCT00568217
Title: Antipyretics for Preventing Recurrences of Febrile Seizures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Heikki Rantala, Professor, University of Oulu, Finland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: fs07hr; K56721
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Last update posted 2007-12-11 (Estimated); Status verified 2007-12

CONDITIONS: Recurrence of Febrile Seizure
MeSH Terms: interventions — Diclofenac; Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 drug (Active Comparator): diclofenac 15 mg/kg suppository once
  Interventions: Drug: Diclofenac, Paracetamol, Ibuprofen
- 2 drug (Placebo Comparator): Placebo suppository once
  Interventions: Drug: Diclofenac, Paracetamol, Ibuprofen
- 3 drug (Active Comparator): acetaminophen mixture 15 mg/kg up to four times a day
  Interventions: Drug: Diclofenac, Paracetamol, Ibuprofen
- 4 drug (Active Comparator): ibuprofen mixture 10 mg/kg up to four times a day
  Interventions: Drug: Diclofenac, Paracetamol, Ibuprofen
- 5 drug (Placebo Comparator): oral placebo mixture up to four times a day
  Interventions: Drug: Diclofenac, Paracetamol, Ibuprofen

INTERVENTIONS:
Drug: Diclofenac, Paracetamol, Ibuprofen — Immediately if temperature > 38 degree Celsius, diclofenac suppository 1,5 mg/kg once or placebo suppository After eight hours, if temperature still < 38 degree Celsius, acetaminophen mixture 15 mg/kg up to four times a day, or ibuprofen mixture 10 mg/kg up to four times a day, or placebo mixture up to four times a day as long as temperature < 38 degree Celsius

SUMMARY:
We wanted to find out if the early use of antipyretics is capable in preventing recurrences of febrile seizures. When a child has had his/her first febrile seizure, the parents were instructed to give him/her antipyretic medication every time when the child had a new episode of fever during two years.

ELIGIBILITY:
Inclusion Criteria:

* First febrile convulsion

Exclusion Criteria:

* Any prior convulsion or antiepileptic medication

Ages: 3 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 231 (Actual)
Dates: Start 1997-09; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
recurrence of febrile seizure | two years

SECONDARY OUTCOMES:
we only had the primary outcome measure | two years

CONTACTS AND LOCATIONS:
Overall Officials: Heikki Rantala, Professor, Principal Investigator — University of Oulu
Locations (1):
- Heikki Rantala, Oulu, Finland

REFERENCES:
- [Derived] Strengell T, Uhari M, Tarkka R, Uusimaa J, Alen R, Lautala P, Rantala H. Antipyretic agents for preventing recurrences of febrile seizures: randomized controlled trial. Arch Pediatr Adolesc Med. 2009 Sep;163(9):799-804. doi: 10.1001/archpediatrics.2009.137. PMID 19736332